CLINICAL TRIAL: NCT06423170
Title: Camrelizumab Plus Gemcitabine and Oxaliplatin (GEMOX) in Patients for Unresectable Gallbladder Cancer: a Single-arm, Phase II Trial
Brief Title: A Single-arm Phase II Clinical Study of the Efficacy and Safety of Camrelizumab Combined With GEMOX for Unresectable GBCs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-516
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Unresectable Gallbladder Cancer
Keywords: PD-1；GEMOX；Unresectable gallbladder cancer.
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus GEMOX (Experimental): Camrelizumab plus GEMOX was given as conversion therapy for unresectable gallbladder cancer
  Interventions: Drug: Camrelizumab plus GEMOX

INTERVENTIONS:
Drug: Camrelizumab plus GEMOX — 1. Camrelizumab：200mg，D1，intravenous infusion, the administration time is 60 (+15) minutes.
  2. GEMOX chemotherapy : oxaliplatin 100mg/m2，D1, gemcitabine1000mg/m2，D1，intravenous infusion.
  3. Carrilizumab and GEMOX chemotherapy will be intravenous infused atone day. Three weeks is a course of treatment,a total of 6-8 courses.

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of Camrelizumab combined with gemcitabine and oxaliplatin (GEMOX) for unresectable gallbladder cancer. Patients with unresectable gallbladder cancer were enrolled to receive gemcitabine 1000mg/m2 D1+oxaliplatin 100mg/m2, D1+Camrelizumab 200mg, D1, in 21-day cycles for 6-8 cycles, with serum tumour markers assessed at each course and abdominal CTA performed every two courses, until tumour progression occurs.The primary indicators of this study are radical tumor resection rate; secondary indicators are disease control rate, objective response rate,progression-free survival and overall survival; safety indicators: incidence and severity of adverse events (AEs) and serious adverse events (SAEs) according to NCI-CTCAEv5.0 criteria. 37 patients are expected to be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years
2. Patients with unresectable gallbladder cancer clearly diagnosed by puncture pathology or the presence of tumour cells in the bile
3. No history of chemotherapy or immunotherapy
4. ECOG score 0-1 within 1 week prior to enrollment
5. Expected survival > 3 months
6. The functional indicators of important organs meet the following requirements： (1)Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; (2)Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range; (3)Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal; (4)Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min(calculated by Cockcroft-Gault formula);
7. Female subjects of childbearing potential must have had a negative serum pregnancy study within 14 days prior to the start of study treatment and be willing to use a reliable method of contraception during the study and for 60 days after the final administration of study drug
8. Male subjects whose partner is a woman of childbearing age should agree to use a reliable method of contraception for the duration of the study and for 120 days after the last dose of study drug
9. Subjects who voluntarily enter the study, sign an informed consent form, are compliant and willing to cooperate with follow-up

Exclusion Criteria:

1. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary carcinoma;
2. Have used gemcitabine-based chemotherapy or have used PD-1 monoclonal antibody or PD-L1 monoclonal antibody treatment within 6 months;
3. Severe cardiopulmonary and renal dysfunction;
4. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2measurements);
5. Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
6. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000;
7. A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment;
8. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period;
9. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive;
10. A history of psychotropic drug abuse, alcohol or drug abuse;
11. Known to have a history of severe allergies to any monoclonal antibodies, platinum drugs, or gemcitabine;
12. Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
radical tumor resection rate | 6 months
  The proportion of patients with negative surgical resection margins in the study group

SECONDARY OUTCOMES:
Disease Control Rate，DCR | 6 months
  The proportion of patients whose tumours shrink or remain stable for a certain period of time and includes cases of complete remission (CR), partial remission (PR) and stable (SD).
Progress Free Survival，PFS | 6 months
  The time between the start of treatment for disease and the observation of disease progression or the occurrence of death from any cause
Overall Survival，OS | 6 months
  The time between the start of the diagnosis of unresectable gallbladder cancerand death from any cause
Objective response rate，ORR | 6 months
  The proportion of patients whose tumour volume shrinks to a pre-defined value and who are able to maintain the minimum time requirement is the sum of the proportion in complete remission (CR) and partial remission (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Rui, PhD, Study Chair — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No